CLINICAL TRIAL: NCT03802305
Title: Comparison of the Variations of the Cardiovascular Parameters and the Efficiency of the Osteocentral Anesthesia (Quicksleeper™) and the Locoregional Anesthesia in the Case of Mandibular Pulpitis
Brief Title: Comparison of Osteocentral Versus Locoregional Anesthesia in Case of Mandibular Molar Pulpitis
Acronym: COQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC18_0268
Record Dates: First submitted 2018-12-19; First posted 2019-01-14 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Endodontic Inflammation
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Intervention Model Description: Number of Arms: 2 Masking: Simple Blinded, Masked Roles: Subject Allocation: Randomized Study Endpoint Classification: Interventional Research with Minimal Risk and Constraints, Safety/Efficacy Enrollment: subjects (anticipated)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized intraosseous technique (Quicksleeper™) (Experimental): patients will receive the anesthetic solution with computerized intraosseous technique anesthesia near the tooth roots involved.
  Interventions: Device: computerized intraosseous technique (Quicksleeper™)
- loco-regional anesthesia (IANB technique) (Active Comparator): patients will receive the anesthetic solution with the loco-regional anesthesia technique: near the place where the nerve goes into the jaw, based on osteo muscular markers.
  Interventions: Device: loco-regional anesthesia (IANB technique)

INTERVENTIONS:
Device: computerized intraosseous technique (Quicksleeper™) — The anesthetic solution is administered with a specific equipment allowing the injection step by step:
  * anesthesia of the interdental papilla,
  * positioning of the needle and perforating of the interdental space,
  * Injection of the solution. All of these steps are based on an adjustment of the different part of this equipment.
  Arms: Computerized intraosseous technique (Quicksleeper™)
Device: loco-regional anesthesia (IANB technique) — The anesthetic solution is delivered by a needle near to the inferior alveolar nerve before it enters the mandibular foramen.
  Arms: loco-regional anesthesia (IANB technique)

SUMMARY:
The irreversible acute pulpitis is the most common emergency at the hospital during dental consultation. Pulpitis are characterized by intense and spontaneous oro-facial pains. In case of mandibular molar, the emergency treatment consists in realizing a pulpotomy (eviction of cameral pulp) under locoregional anesthesia called inferior alveolar nerve block (IANB). The latter represents a real challenge, since inflammation may decrease its action. To mitigate this deficiency and the drawbacks of the IANB (onset and duration of the anesthesia, bites risk reported with IANB) other anesthesias are proposed. In particular the computerized intraosseous technique anesthesia of which the Quicksleeper™ system is a part. However, according to the observers, a mild to severe tachycardia have been reported.

Very few valid clinical trials exists on the subject, most being realized with systems of intraosseous anesthesia other than Quicksleeper™. Therefore, the aim of this study is first to analyze the variations of the cardiovascular parameters into two groups of anesthesia: locoregional anesthesia and Quicksleeper ™ system; and then, to compare the efficiency, side effects, operating consequences of both techniques. This study should provide better data about potential risk with computerized intraosseous technique such has Quicksleeper ™ system in healthy or cardiovascular risk patient.

DETAILED DESCRIPTION:
When the patient arrive in the dental care center, an initial assessment is made to get the diagnosis of irreversible pulpitis:

1. Anamnesis:

   acute and spontaneous oro-facial pain, pulsatile severe intensity, which could irradiate toward the ear and/or jaw, exacerbated by cold or hot.
2. Clinical exams: positive vitality tests (electric test and cold pressor test)
3. Further examination (radiography)

The inclusion and exclusion criteria will be checked and the informed consent of the patient will be taken. The patient is then randomized in one of the group (experimental or control). He will fill a questionnaire (Corah's scale) for evaluating his state of anxiety during care. A monitoring of cardiac parameters is made during the care at defined moment.

The patient evaluates his pain himself with the VAS (Visual Analog Score), before the intervention. The anesthesia is carried out by only one experimenter, with the Quickslepper™ handpiece but different specific needles.

Each patient receive 1.8 mL of 4% articaine 1:100 000 on a period of 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* real irreversible pulpitis of a mandibular molar in dental emergency consultation at the Nantes hospital
* Healthy patient without medical history (ASA 1), without treatment for heart rate distress (anti arrhythmic, beta-blocking drug)
* Major and covered by the social security
* Informed consent

Exclusion Criteria:

* ASA > 1
* Pregnant and breastfeeding women
* Minors
* Adults under guardianships
* Adults deprived of freedom
* Impossibility to obtain for informed consent
* Allergy to anesthetic components
* Contraindication of vasoconstrictor
* Angle closure glaucoma

  * Pheochromocytomas
  * Bisphosphonate IV
  * Irradiated patient (upper respiratory and gastrointestinal tract cancer)
  * Contraindication with Mono-amino oxidase inhibitors
* Acute apical periodontitis
* Pulpitis on wisdom teeth
* Vital teeth with fixed prosthesis
* Active periodontal disease
* Local anatomic difficulty
* No reference tooth for vitality dental test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
time required (in minutes) to re-obtain the baseline cardiovascular parameters like reported before injection: expected event. | at day 0, from T0 minute to T14 minutes
  * 3 successive values of heart rate similar to those registered before injection.
  * 3 successive values of blood pressure (diastolic and systolic) similar to those registered before injection.

SECONDARY OUTCOMES:
Compare the pain of the patient between the two anesthetic techniques | 3 days
  Scores measured with Visual Analog Score( Heft-Parker's pain assessment) (minimum score : no pain ; maximal score : maximum pain unimaginable)
Compare the possible postoperative course between the 2 anesthetic techniques | 3 days
  The postoperative course will be evaluated using a post-operative table to be completed by the patient at Day + 1, Day + 2 and Day + 3. Collection of information by phone call to the patient. The presence or absence of the following item is measured : pain after waking up, swelling, hematoma, seepage, higher tooth sensation, bite, possibility of feeding, mouth opening limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes Universitary Hospital, Nantes, Loire-Atlantique, France

REFERENCES:
- [Derived] Gaudin A, Clouet R, Boeffard C, Laham A, Martin H, Amador Del Valle G, Enkel B, Prud'homme T. Comparing intraosseous computerized anaesthesia with inferior alveolar nerve block in the treatment of symptomatic irreversible pulpitis: A randomized controlled trial. Int Endod J. 2023 Aug;56(8):922-931. doi: 10.1111/iej.13935. Epub 2023 May 29. PMID 37209243
- [Derived] Laham A, Clouet R, Del Valle GA, Gaudin A, Prud'homme T. Anaesthetic efficacy and influence on cardiovascular parameters change of intraosseous computerised anaesthesia versus inferior alveolar nerve block anaesthesia in acute irreversible pulpitis of mandibular molars: study protocol for a prospective randomised controlled trial. Trials. 2022 Dec 5;23(1):979. doi: 10.1186/s13063-022-06915-4. PMID 36471427